CLINICAL TRIAL: NCT00920166
Title: Growth and Tolerance in New Born Fed Formula Supplemented With Alpha-Lactalbumin and Containing a Symbiotic
Brief Title: Evaluation of Safety, Growth, Tolerance and Effects on the Intestinal Fora of a New Milk for Healthy Infants
Acronym: Pétunia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sodilac (Industry)
Responsible Party: Pr Jean Christophe Rozé (Principal investigator), CHU de Nantes
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: PET-CL3-001
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Growth
Keywords: Infant formula; Alpha-lactalbumin; Symbiotic; Allergy; Gastrointestinal tolerance; Bacterial colonization; Faecal IgA analysis
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modilac Pétunia 1 (Experimental): Formula with reduced total protein concentration, enriched in alpha-lactalbumin and containing a symbiotic
  Interventions: Dietary Supplement: Pétunia 1
- Modilac 1 (Active Comparator): Regular milk
  Interventions: Dietary Supplement: Regular formula

INTERVENTIONS:
Dietary Supplement: Pétunia 1 — Infant formula used for non breastfed children
  Other Names: Modilac Pétunia 1
  Arms: Modilac Pétunia 1
Dietary Supplement: Regular formula — Infant formula used for non breastfed children
  Other Names: Modilac 1
  Arms: Modilac 1

SUMMARY:
The purpose of the study is to assess growth and tolerance in new born and infant fed an experimental infant formula with reduced total protein concentration, enriched in alpha-lactalbumin and containing a symbiotic.

DETAILED DESCRIPTION:
This prospective, randomized, double blind, controlled study evaluated the safety and effect on growth and tolerance to an infant formula supplemented with alpha-lactalbumin and containing a symbiotic, in term infants.

Term infants with a gestational age ranging from 37 to 42 weeks and whose parents chose formula feeding were enrolled during their first eight days of life.

Both parents provided informed written consent. Infants were randomly assigned to receive either the new test formula or a control, a regular formula adapted for term infants (Modilac®1). The control formula is formulated to meet the nutritional needs of infants.

For each neonates, neonatal parameters were collected.

5 visits took place : V1 (inclusion), V2 (randomization), V3 (1 month), V4 (3 months) and V5 (6 months). During each visit, the investigator filled in observational book the anthropometric parameters (weight, height, head circumference, BMI) and pieces of information collected 3 days before by the parents (gastrointestinal tolerance parameters, daily infant behaviour and milk consumption). Global parents' contentment was evaluated as well.

In two investigation centers, at the end of the 6th month, immuno-allergic test was realised.

Stools were collected at the end of the first and sixth month from diapers, for microbiological analysis and measurements of faecal inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Term health newborn infant with gestational age ranging from 37 to 42 weeks
* Eutrophic
* Non breastfed children
* Apgar score > 5 to 7 minutes

Exclusion Criteria:

* Infant presenting a metabolic, nervous, digestive or organic disease able to interfere with study
* Evidence of protein cow milk allergy
* Infant presenting lactose intolerance
* Newborn whose parents did not provide informed consent
* Newborn currently participating in another trial

Max Age: 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Growth Parameters | 1, 3 and 6 months

SECONDARY OUTCOMES:
Sensitization or allergy | 1, 3 and 6 months
Atopic diseases (eczema atopic, asthma, allergic rhinitis) | 1, 3 and 6 months
Describe the intestinal flora according to the nutrition group | 1 and 6 months
Clinical Tolerance | 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe Rozé, PhD, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - CHU d'Angers, Angers
  - CHU de Nantes, Nantes
  - Hôpital Saint Vincent de Paul (AP-HP), Paris
  - Hôpital de la Pitié Salpétrière, Paris

REFERENCES:
- [Derived] Roze JC, Barbarot S, Butel MJ, Kapel N, Waligora-Dupriet AJ, De Montgolfier I, Leblanc M, Godon N, Soulaines P, Darmaun D, Rivero M, Dupont C. An alpha-lactalbumin-enriched and symbiotic-supplemented v. a standard infant formula: a multicentre, double-blind, randomised trial. Br J Nutr. 2012 Jun;107(11):1616-22. doi: 10.1017/S000711451100479X. Epub 2011 Nov 14. PMID 22079177